CLINICAL TRIAL: NCT04289480
Title: ENTERPRISE 2 Vascular Reconstruction Device and Delivery System Registry: A Multicenter, Prospective, Single-arm Observational Study to Evaluate the Safety and Effectiveness With the Device to Facilitate Endovascular Coil Embolization of Intracranial Aneurysms
Brief Title: Safety and Effectiveness of ENTERPRISE 2 Device in the Endovascular Treatment of Intracranial Aneurysms
Acronym: EMPOWER
Status: Active, not recruiting | Type: Observational
Sponsor: Medos International SARL (Industry)
Collaborators: Johnson & Johnson Medical (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNV_2018_02
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial aneurysms, Neurovascular
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ENTERPRISE 2 group: The study population enrolled for this clinical study is "aneurysm patients who need stent-assisted coiling treatment", using ENTERPRISE 2 device.
  Interventions: Device: ENTERPRISE 2 device

INTERVENTIONS:
Device: ENTERPRISE 2 device — The ENTERPRISE 2 Vascular Reconstruction Device is intended for use with occlusive devices in the treatment of intracranial aneurysms.

SUMMARY:
The study is designed to evaluate the safety and effectiveness of ENTERPRISE 2 vascular reconstruction device and delivery system (hereinafter referred to as ENTERPRISE 2) to facilitate endovascular coil embolization of intracranial aneurysms.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm observational study, in which enrolled patients will be implanted with the ENTERPRISE 2 for evaluation of safety and effectiveness of ENTERPRISE 2 in real-world applications.

The study population will consist of 164 patients with ruptured or unruptured intracranial aneurysms and a parent vessel diameter of ≥2.5 mm and ≤4 mm. All patients will be implanted with the study device.

The enrolled patients will be followed at 30 days, 180 days, 1 year, 2 years, 3 years, 4 years and 5 years post procedure.

The primary endpoint is the incidence of aneurysm recanalization (at 180 days) evaluated through digital subtraction angiography (DSA). Secondary effectiveness endpoints include incidence of aneurysm recanalization (at 1 year), successful stent/coil placement rate (immediately post procedure), aneurysm occlusion (immediately post procedure, at 180 days and 1 year), incidence of retreatment (at 30 and 180 days, and 1, 2, 3, 4 and 5 years). Safety evaluation include: incidence of disabling stroke or neurological death (at 180 days and 1 year), incidence of in-stent thrombosis (at 180 days and 1 year), and incidence of in-stent stenosis (at 180 days and 1 year). Exploratory endpoints include stent wall apposition performance (intra-procedure), first-time deployment success rate (intra-procedure) and duration of stent deployment (intra-procedure).

ELIGIBILITY:
Inclusion Criteria:

1. Patient (or his/her legal representative) understands the nature of the procedure and provides voluntary written informed consent for the use of his/her peri-procedural and follow-up data;
2. Aged between 18 years and 80 years of age the time of consent;
3. Patient has been diagnosed with ruptured (Hunt-Hess Grade I-III) or unruptured intracranial aneurysm and requires the endovascular treatment;
4. Parent vessel with a diameter of ≥2.5 mm and ≤4 mm;
5. Patient is willing to return to the investigational site for the post-procedure follow-up evaluations.

Exclusion Criteria:

1. Severe co-morbidity associated with a life-expectancy of less than twelve months as determined by the investigator;
2. Poor clinical condition with modified Rankin Scale (mRS) score ≥4;
3. Having prior or potential severe allergic reaction to contrast medium;
4. Known allergies to any of the device components, including Enterprise 2 and PROWLER® SELECT™ Plus Infusion Catheter;
5. Angiogram demonstrating that the aneurysm is not appropriate for endovascular treatment (i.e. severe intracranial vessel tortuosity, stenosis, intracranial vasospasm not responsive to medical therapy);
6. Arteriovenous malformation (AVM) in the territory of the target aneurysm;
7. Unsuitable for the antithrombotic and/or anticoagulant therapies;
8. Implantation of an intracranial stent associated with aneurysm or symptom distribution within 12 weeks prior to signature of Informed Consent Form;
9. Implantation of a carotid stent associated with aneurysm or symptom distribution within 12 weeks prior to signature of Informed Consent Form;
10. Evidence of active infection;
11. Pregnant or lactating women;
12. Having participated in clinical studies of other investigational drugs or devices within 30 days prior to signature of Informed Consent Form, excluding epidemiological studies of observational nature or natural history or not involving intervention;
13. Pre-planned staged procedure of target aneurysms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in patients with unruptured or ruptured intracranial aneurysm with a parent vessel diameter of ≥2.5 mm and ≤4 mm.
Sampling Method: Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of aneurysm recanalization | at 180 days post procedure
  Incidence of aneurysm recanalization (at 180 days) = number of target aneurysm recanalization (at 180 days) ÷ total number of target aneurysms receiving follow-up × 100%. The results of aneurysm angiography at 180-day follow-up will be obtained through DSA, and the post-procedure immediate aneurysm recanalization shown in angiograms will be graded as per the Raymond-Roy Classification Scale.
  The Raymond-Roy Classification at each follow-up time point increased by ≥ one class relative to that immediately after the procedure is defined as recanalization (e.g., Class I immediately after the procedure, Class II at 180-day follow-up).

SECONDARY OUTCOMES:
Incidence of aneurysm recanalization | at 1 year post procedure
  Incidence of aneurysm recanalization (at 1 year) = number of target aneurysm recanalization (at 1 year) ÷ total number of target aneurysms receiving follow-up × 100%. The results of aneurysm angiography at 1 year follow-ups will be obtained through DSA or MRA or CTA.
Successful stent/coil placement rate | immediately post procedure
  Successful stent/coil placement rate = number of target aneurysms with successful stent/coil placement ÷ total number of target aneurysms× 100%.
  Successful stent/coil placement is defined as successful stent deployment and successful delivery and placement of the coil at the target aneurysm assessed immediately post procedure through angiography.
Aneurysm occlusion | immediately post procedure, at 180 days and at 1 year post procedure
  Aneurysm occlusion rate = number of target aneurysms with Raymond-Roy Class I or II aneurysm occlusion÷ total number of target aneurysms× 100%.
  The aneurysm occlusion will be assessed by classifying the post-procedure immediate aneurysm occlusion shown in angiograms based on the Raymond-Roy Classification.
Incidence of retreatment | at 30 days, 180 days, 1 year, 2 years, 3 years, 4 years and 5 years post procedure
  Incidence of retreatment = number of target aneurysms receiving retreatment during the follow-up ÷ total number of target aneurysms receiving follow-up ×100%.
  Retreatment refers to any intervention to the target aneurysm after completing first stent-assisted coil embolization for the target aneurysm.

OTHER OUTCOMES:
Incidence of disabling stroke or neurological death | at 180 days, at 1 year post procedure
  Incidence of disabling stroke or neurological death = number of patients with disabling stroke or neurological death ÷ total number of patients receiving follow-up × 100%.
  Stroke is defined as rapidly developing clinical signs of focal (or global) disturbance of cerebral function lasting more than 24 hours with no apparent cause other than of vascular origin, including ischemic stroke or hemorrhagic stroke (i.e., intraparenchymal hemorrhage (IPH), SAH, subdural hemorrhage (SDH), epidural hemorrhage (EDH)).
  Disabling stroke is defined as mRS score ≥ 3 assessed at a minimum of 90 days (+/- 30 days) post-stroke event.
  Neurological death, also called brain death, refers to irreversible loss of the capacity for consciousness combined with the irreversible loss of all brainstem functions, including the capacity to breathe.
Incidence of in-stent thrombosis | at 180 days, at 1 year post procedure
  Incidence of in-stent thrombosis = number of target aneurysms with parent vessel (in-stent) thrombosis during follow-up ÷ total number of target aneurysms receiving follow-up ×100%.
Incidence of in-stent stenosis | at 180 days, at 1 year post procedure
  Incidence of in-stent stenosis = number of target aneurysms with parent vessel (in-stent) stenosis during follow-up ÷ total number of target aneurysms receiving follow-up ×100%.
  Mild, moderate, and severe in-stent stenosis is clinically defined as a stenosis of <33%, 33-67%, and ≥67%, respectively, comparing with non-stented parent vessel [43, 44]. In this study, moderate and severe in-stent stenoses (with a stenosis of ≥33%) of the parent vessel are defined as in-stent stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Xinjian Yang, Professor, Principal Investigator — Beijing Tiantan Hospital; Shiqing Mu, Professor, Principal Investigator — Beijing Tiantan Hospital; Qingrong Zhang, Professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Yuxiang Gu, Professor, Principal Investigator — Huashan Hospital Shanghai Medical college, Fudan University; Chuanzhi Duan, Professor, Principal Investigator — Southern Medical University, China; Shu Wan, Professor, Principal Investigator — Zhejiang Hospital; Bo Yu, Professor, Principal Investigator — Shengjing Hospital; Yang Wang, Professor, Principal Investigator — The First Affiliated Hospital of Nanchang University; Sheng Guan, Professor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Wohua Zhao, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science & Technology; Xinjian Yang, Professor, Principal Investigator — Beijing Anzhen Hospital
Locations (10):
- China (10):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The first affiliated hospital of Nanchang university, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Huashan Hospital Shanghai Medical college, Fudan University, Shanghai, Shanghai Municipality
  - Zhejiang Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.